CLINICAL TRIAL: NCT04436432
Title: Phenomenology of Anxiety in Preschool Children With Autism Spectrum Disorder
Brief Title: Phenomenology of Anxiety in Preschool Children With ASD
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Roma Vasa, Director of Psychiatric Services, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: IRB00173329
Record Dates: First submitted 2020-06-04; First posted 2020-06-18 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Anxiety; Autism Spectrum Disorder
Keywords: Autism; Anxiety; Eye tracking; Preschool
MeSH Terms: conditions — Anxiety Disorders; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment: Children with ASD ages 3-5 years at baseline

SUMMARY:
This study investigates the prevalence, phenomenology, and correlates of anxiety in preschool children with autism spectrum disorder (ASD) across a two-year period. Attention bias to threat, a potential objective marker of anxiety, also is examined using eye tracking methods.

DETAILED DESCRIPTION:
Anxiety disorders in children with autism spectrum disorders (ASD) are one of the most prevalent and impairing co-occurring conditions, affecting approximately 40% of the population and causing major disruptions in school and family life. Research in typically developing (TD) children suggests that anxiety usually emerges in the preschool years (3-5 years) and can result in future psychopathology. Early detection and treatment of childhood anxiety in children with ASD can lead to improved clinical outcomes.

This study assesses the prevalence and phenomenology of anxiety in preschool children with ASD utilizing an established and comprehensive measure of anxiety in children with ASD across three time points (baseline, one year post, two years post).It also investigates the association of child (e.g., ASD features) and parent (e.g., mental health, caregiver strain) characteristics with anxiety cross-sectionally and longitudinally, to determine if certain correlates predict or maintain future anxiety. Attention bias to threat stimuli and its physiological correlates are also examined as potential objective markers of anxiety using eye tracking and pupillometry methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 years 0 months to 5 years 11 months;
* DSM-5 ASD diagnosis based on clinical impressions and results of the Autism Diagnostic Observation Schedule-2 (ADOS-2)
* Child resides with at least one biological parent
* Parents are English speaking

Exclusion Criteria:

* History of psychological trauma
* History of neurologic illness
* Parent substance abuse, bipolar disorder, psychosis
* Parents require support from a medical interpreter
* Child displays severe behavior challenges
* Severe eyesight or hearing impairments that may interfere with the protocols

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Clinical and community based sample
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Anxiety diagnostic status as measured by Anxiety Disorders Interview Schedule with Autism Addendum | Anxiety diagnostic status will be measured through study completion, up to 24 months
  Gold-standard semi-structured interview for assessing anxiety disorders and the ASA, a supplement to the ADIS that facilitates the use of this tool in children with ASD; clinical severity ratings range from 0 to 3 or 0 to 8; higher scores indicate more impairment
Attention to threat behavioral paradigms | Attention to threat and correlated physiological arousal will be measured across the final 12 months of the study
  Child's attention to threatening stimuli measured via eye tracking and correlated physiological response measures via pupillometry; more frequent saccades to threatening stimuli indicate higher attention bias to threat; greater pupil dilation indicates higher physiological arousal

SECONDARY OUTCOMES:
Child Behavior Checklist | Anxiety and other psychiatric symptoms will be assessed through study completion, up to 24 months
  parent and teacher report scale that measures child anxiety and other psychiatric symptoms;T scores range from 20 to 100; Syndrome scales: T-scores over 65 indicate clinically significant symptoms
Preschool Anxiety Scale - Revised | Anxiety will be assessed through study completion, up to 24 months
  parent and teacher report scale measuring levels of anxiety in preschool aged children; scores range from 0 to 112; higher scores indicate higher anxiety
Screen for Child Anxiety Related Disorders | Anxiety will be assessed through study completion, up to 24 months
  parent and teacher report scale measuring levels of anxiety in children 6 or older; scores range from 0 to 114; higher scores indicate higher anxiety
Response to Uncertainty and Low Environmental Stability Scale | Intolerance of uncertainty will be assessed through study completion, up to 24 months
  parent and teacher report scale measuring response to uncertainty and low environmental structure in children; scores range from 1 to 5; higher scores indicate higher intolerance of uncertainty
Social Responsiveness Scale | ASD symptoms will be assessed through study completion, up to 24 months
  parent report scale that assesses the presence and severity of social impairment in children; T-scores range from 20 to 100; higher scores indicate higher ASD severity
Emotion Regulation Checklist | Emotional regulation will be assessed through study completion, up to 24 months
  parent report scale that assesses emotion regulation capacities in children; scores range from 24 to 96; higher scores indicate higher impairment
The Children's Sleep Habits Questionnaire | Sleep habits will be assessed across the final 12 months of the study
  parent report questionnaire that measures sleep habits in children; scores range from 45 to 135; higher scores indicate greater frequency of sleep problems
Hospital Anxiety and Depression scale | Parental anxiety and depression will be assessed through the completion of the study, up to 24 months
  screening tool that will be used to capture clinical anxiety and depression in parents; scores range from 0 to 21; higher scores indicate higher anxiety and/or depression symptoms
Intolerance of Uncertainty Scale | Parental intolerance of uncertainty will be assessed through the completion of the study, up to 24 months
  scale that will be used to measure parental responses to uncertainty, ambiguous situations and the future; scores range from 12 to 60; higher scores indicate higher intolerance of uncertainty
Family Accommodation Scale | Parental accommodation will be assessed through the completion of the study, up to 24 months
  assesses parental accommodation of child's interfering symptoms; scores range from 0 to 36; higher scores indicate higher parental accommodation
Burden Assessment Scale | Parental strain will be assessed through study completion, up to 24 months
  measures strain (thoughts, feelings, disruption) associated with having a child with a neurodevelopmental disorder; scores range from 19 to 76; higher scores indicate greater family burden
Broader Autism Phenotype | Parental autism features will be assessed through study completion, up to 24 months
  self-report scale that measures broader autism symptoms in the parent; scores range from 36 to 216; higher scores indicate greater severity of autism features

CONTACTS AND LOCATIONS:
Overall Officials: Roma A Vasa, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasa RA, Kreiser NL, Keefer A, Singh V, Mostofsky SH. Relationships between autism spectrum disorder and intolerance of uncertainty. Autism Res. 2018 Apr;11(4):636-644. doi: 10.1002/aur.1916. Epub 2018 Jan 7. PMID 29316350
- [Background] Vasa RA, Keefer A, Reaven J, South M, White SW. Priorities for Advancing Research on Youth with Autism Spectrum Disorder and Co-occurring Anxiety. J Autism Dev Disord. 2018 Mar;48(3):925-934. doi: 10.1007/s10803-017-3320-0. PMID 29164436
- See also: Study Flier — https://www.kennedykrieger.org/sites/default/files/library/documents/patient-care/centers-and-programs/center-for-autism-and-related-disorders/FINAL_IRB00173329_Study%20flyer_revised%20(1).pdf